CLINICAL TRIAL: NCT04154878
Title: Novel Echo Diastolic Measurements (Index)
Brief Title: 2 New Measurements Used to Describe the Filling Phase of the Left Ventricle (LV).
Acronym: INDEX
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1384494
Record Dates: First submitted 2019-10-31; First posted 2019-11-07 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Diastolic Heart Failure; Left Ventricular Diastolic Dysfunction; Left Ventricular Diastolic Collapse
MeSH Terms: conditions — Heart Failure, Diastolic; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pacemaker Optimization: Participants were referred for pacemaker optimization following implantation of a device. All had an intact atrial contraction either intrinsic or by device stimulation. A standard baseline echo was performed prior to programming changes with a final echo scan completed after all programming complete. Device programming consisted of adjusting atrial ventricular and right to left ventricular stimulation delays.
- Healthy: A brief cardiac history questionnaire and complete echocardiogram will be performed.

SUMMARY:
As we live longer our population experiencing heart failure (HF) continues to grow consuming an increasing percent of healthcare dollars. Systolic heart failure or pump failure is easy to recognize and measure and is expressed as ejection fraction. Diastolic heart failure (DHF) or failure to fill adequately is much more difficult to quantify with no single measure or number being used to express the severity instead groupings are used with normal and Grade I, II or Grade III to classify with Grade III being the direst.

Heart Failure with Reduced Ejection Fraction (HFrEF) and Heart Failure with Preserved Ejection Fraction (HFpEF) are used to identify the primary clinical presentation of HF but do not adequately describe the combined effect often presenting within the same subject. It is estimated 35 to 50% of those with HFrEF, having Left Ventricle Ejection Fraction (LVEF) < 50%, and 50 to 70% of those with HFpEF, having ejection fraction ≥ 50%, also have moderate to severe diastolic dysfunction (DD).

The purpose of this study is two fold. The first is to determine if the rate of change measured from the left ventricular inflow inspiratory phase Doppler waveform provides insight into a cause of diastolic heart failure by comparing echocardiographic data points obtained prior to and immediately following optimization of a bi-ventricular pacemaker. This HF population requires an ejection fraction of 35 percent or lower to qualify for the device. These echocardiograms have been previously completed and will be reanalyzed.

The second purpose is to determine if relationships between different features of a LV volume curve can be used to generate a single number to describe global diastolic function using the same echocardiograms from the pacemaker group.

Results will be compared to a small group of healthy normal participants as a control for validation.

DETAILED DESCRIPTION:
The purpose of this study is to introduce novel measurements to improve the classification of ventricular diastolic performance.

There are 2 cohorts. Cohort 1 consists of 100 subjects who were referred and received echo guided biventricular pacemaker optimization. This retrospective component data is being retrieved to compare baseline and final cardiac performance measures. Comparisons will be made between Doppler and 3D echo diastolic and systolic markers. The Doppler diastolic markers will include D-E slope measuring the rate of pressure equalization between the left atrium (LA) and left ventricle (LV) during inspiration and expiration. MV VTI, the velocity time integral of the left ventricular inflow tract (LVIT) a surrogate measure for LV filling volume, averaging three consecutive complexes and minimal and maximal variability. TDI, tissue Doppler Imaging, when coupled with LVIT measures provides an estimation of left ventricular diastolic pressure. IRT, isovolemic relaxation time, an indicator of LA preload, S/D ratio, an indicator of LA compliance/pressure compared to pulmonary venous pressure. LAv, LA volume, a criteria for diastolic dysfunction grading. TRvmax, tricuspid regurgitation maximum velocity, used to estimate right ventricular systolic pressure. 3D measures will be obtained from the volume curve generated from the 3D full volume image acquisition. The 2 slopes being compared are the initial filling (R1) and intermediate filling (R2) rates of volume change over time or R1/R2. LV ejection fraction, diastolic filling time (DFT), ejection time (ET), heart rate (HR), initial filling time (IFT), and stroke volume (SV) are all being measured from the 3D volume curve.

Cohort 2 consists of normal healthy participants to serve as a comparison providing HF diseased state differentiation. All baseline measures performed in cohort 1 will be done for cohort 2.

Primary Objective/Aim/Goal/Hypothesis Hypothesis: To determine if LV volume curves can be used to generate a single number that globally describes diastolic function and identify relationship to current grouping algorithm.

Secondary Objective/Aim/Goal/Hypothesis Hypothesis: To determine if the pulse wave Doppler of the left ventricular inflow tract D-E slope measure and changes correlate with changes in diastolic performance of the LV.

Hypothesis: Does weighting of the volume curve analysis with various features of the curve such as stroke volume, initial filling volume, and initial filling volume percent provide greater sensitivity or specificity in differentiating diastolic performance.

Study Design: This study is a retrospective observational data analysis of echocardiographic images and Doppler waveforms comparing data between measurements and calculations taken at baseline and after final programming of biventricular pacemaker devices performed during a single visit. Additionally, the echo data from 5 normal healthy participants will be acquired during a single visit to establish normal values and demonstrate reproducibility.

ELIGIBILITY:
Cohort 1

Inclusion Criteria:

1. Underwent pacemaker optimization at study location.
2. Pacemaker optimization between May 1, 2007 and August 16, 2015.
3. Heart rate less than 95 beats per minute.

Exclusion Criteria:

1. Missing Data Points.
2. Poor quality echo images.
3. Atrial fibrillation.

Cohort 2 Inclusion Criteria.

1. Considered in good cardiac condition.
2. Heart rate less than 90 beats per minute.

Exclusion Criteria

History of or treatment for:

1. Atrial fibrillation.
2. Coronary artery disease.
3. Heart Attack.
4. Pacemaker.
5. Cardiomyopathy.
6. Diabetes.
7. Kidney disease.
8. Hypertension. Systolic pressure > 140. Diastolic pressure > 90.
9. Lung disease.
10. Emphysema.
11. Bronchitis.
12. Asthma.

Withdrawal Criteria:

1. Poor quality echo images.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1 participants are individuals who have received a baseline and final echocardiogram.
  Cohort 2 is comprised of cardiac healthy participants.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
LV Volume Curve Classification | 9 months
  Determine the LV Volume Classification based on the current American Society of Echocardiography classification method
D-E Slope | 6 months
  Determine if the D-E Slope contributed additional information to diastolic function classification

SECONDARY OUTCOMES:
LV Volume Curve Weighting of R1/R2 with SV, ET, IFV, DFT | 9 months
  Determine if the use of various volume curve features improve sensitivity
LV Volume Curve Weighting of R1/R2 with body mass indexed SV and IFV | 9 months
  Determine if the use of various volume curve features improve sensitivity
D-E Slope variability comparing minimum and maximum values measured during resting respirations | 9 months
  Is resting D-E Slope variability comparing minimum and maximum values measured during resting respirations associated with diastolic dysfunction severity

CONTACTS AND LOCATIONS:
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagueh SF, Appleton CP, Gillebert TC, Marino PN, Oh JK, Smiseth OA, Waggoner AD, Flachskampf FA, Pellikka PA, Evangelista A. Recommendations for the evaluation of left ventricular diastolic function by echocardiography. J Am Soc Echocardiogr. 2009 Feb;22(2):107-33. doi: 10.1016/j.echo.2008.11.023. No abstract available. PMID 19187853
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Background] Oh JK, Park SJ, Nagueh SF. Established and novel clinical applications of diastolic function assessment by echocardiography. Circ Cardiovasc Imaging. 2011 Jul;4(4):444-55. doi: 10.1161/CIRCIMAGING.110.961623. No abstract available. PMID 21772012
- [Background] 4. Richard J. Moro, US Patent Application Publication US 2014/0275976 A1, Sep 18, 2014